CLINICAL TRIAL: NCT04951570
Title: Clinical Diagnosis and Treatment of Intracerebral Hemorrhage Based on Artificial
Brief Title: Clinical Diagnosis and Treatment of Intracerebral Hemorrhage Based on Artificial Intelligence
Acronym: CATCH-AI
Status: Completed | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Xingquan Zhao, Professor of Neurology and Stroke Center, Beijing Tiantan Hospital
Other Study IDs: CATCH-AI
Record Dates: First submitted 2021-06-20; First posted 2021-07-07 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Intracerebral Hemorrhage
Keywords: Intracerebral Hemorrhage; Hematoma Expansion; Artificial Intelligence
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — blood samples and urine samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hematoma Expansion (HE) group
- non-HE group

SUMMARY:
The purpose of this study is to test the reliability and validity of an artificial intelligence system and a related 5-score scale to predict hematoma expansion, and conduct a study cohort of intracerebral hemorrhage to screen out imaging and biological markers that could predict hematoma expansion in real-world.

DETAILED DESCRIPTION:
This is a investigator-initiated, multi-center, prospective, registered cohort study. The study is intended to enroll 4000 patients with intracerebral hemorrhage from 50 hospital in China. Clinical and imaging data, as well as the results of laboratory examination will be collected to test the reliability and validity of an artificial intelligence system and a related 5-score scale to predict hematoma expansion, and conduct a study cohort of intracerebral hemorrhage to screen out imaging and biological markers that could predict hematoma expansion in real-world.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of spontaneous intracerebral hemorrhage(sICH)
2. Age ≥18;
3. Admission within 24 hours of symptom onset
4. CT available at 24 hours
5. Informed consent obtained

Exclusion Criteria:

1. Intracerebral hemorrhage caused by tumor, vascular malformation, aneurysm, etc.
2. Deep coma at admission (GCS≤8)
3. Intended to have a surgery within 24 hours
4. Congenital coagulation dysfunction
5. Previous intracerebral hematoma have not been absorbed

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with sICH that arrived at hospital within 24 hours.
Sampling Method: Probability Sample
Enrollment: 1374 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
hematoma expansion | 24-48 hours from symptom onset
  non-contrast CT scan: the enlargement of hematoma ≥6ml
Recurrence of intracerebral hemorrhage | 90 days from symptom onset
  non-contrast CT scan: non-traumatic intracerebral hemorrhage other than the primary hemotoma
Functional dependence | 3 months
  modified Rankin Scale score ≥3 (a global measure of disability on a seven-level scale, with scores ranging from 0 (no symptoms) to 6 (death), higher scores mean a better or worse outcome )
Cerebrovascular death | 3 months
  Death due to one of the following events: ischemic stroke or hemorrhagic stroke
Cardiovascular death | 3 months
  Death due to one of the following events: sudden cardiac death or acute myocardial infarction or heart failure

SECONDARY OUTCOMES:
New ischemic stroke | 3 months
  Acute focal neurological impairment corresponding with infarction on CT/MR scan
New subarachnoid hemorrhage | 3 months
  Hemorrhage in subarachnoid space proven on CT/MR scan
Other cardiovascular events | 3 months
  One of the following events: non-fatal myocardial infarction or non-fatal heart failure

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, China